CLINICAL TRIAL: NCT01882543
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of AQX-1125 in Subjects With Interstitial Cystitis/Bladder Pain Syndrome Mediated by the Src Homology-2-domain-containing Inositol 5' Phosphatase [SHIP1] Pathway
Brief Title: Efficacy and Safety of AQX-1125 in IC/BPS
Acronym: LEADERSHIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aquinox Pharmaceuticals (Canada) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AQX-1125-201
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Interstitial cystitis; Bladder pain syndrome; IC/BPS; AQX-1125; SHIP1
MeSH Terms: conditions — Cystitis, Interstitial | interventions — 4-(4-(aminomethyl)-7a-methyl-1-methylideneoctahydro-1H-inden-5-yl)-3-(hydroxymethyl)-4-methylcyclohexan-1-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AQX-1125 (Experimental): 1 x AQX-1125 Capsule daily
  Interventions: Drug: AQX-1125
- Placebo (Placebo Comparator): 1 x placebo capsule daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AQX-1125 — Synthetic SHIP1 activator
  Arms: AQX-1125
Drug: Placebo — Double blind placebo capsule
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of 6 weeks of treatment with once daily administration of AQX-1125 compared to placebo on average daily pain in subjects with interstitial cystitis/bladder pain syndrome (IC/BPS), during and after treatment, using a standardized 11-point numerical rating scale (NRS) pain score recorded by electronic diary

ELIGIBILITY:
Inclusion Criteria:

* Be females, ≥18 and ≤75 years of age, who have consistently had symptoms of bladder pain in addition to urinary urgency and/or urinary frequency for more than 12 months
* Have had the diagnosis of interstitial cystitis for > 6 months (pain for at least 12 months) but ≤15 years
* Have average daily pain score of at least 5 out of 10 on the 11-point Numerical Rating Scale [NRS] pain scale in the 9 days prior to baseline
* Have undergone a cystoscopy and have documented visible signs of bladder bleeding, lesions or glomerulation within the last 36 months prior to baseline.
* Subjects if of child bearing potential, must agree to avoid pregnancy and use medically acceptable method of contraception from screening visit and throughout the study.
* Must be capable of voiding independently

Exclusion Criteria:

* Pelvic floor pain (>5 out of 10 on the 11-point NRS pain scale following a pelvic pain assessment)
* Have a body mass index [BMI] of <18 kg/m2 or >39 kg/m2
* Have had a urinary tract infection including bacterial cystitis within the past 30 days.
* Have greater than 1+ hematuria on dipstick test at screening from an unknown cause
* History of previous procedure(s) (augmentation cystoplasty, cystectomy, or cystolysis) that has affected bladder function

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Shrewsbury, MD, Study Director — Aquinox Pharmaceuticals (Canada) Inc.
Locations (29):
- United States (12):
  - AQX/CMX site, Homewood, Alabama
  - AQX/CMX site, Glendora, California
  - AQX/CMX site, San Diego, California
  - AQX/CMX site, Denver, Colorado
  - AQX/CMX site, Farmington, Connecticut
  - AQX/CMX site, Orlando, Florida
  - AQX/CMX site, Shreveport, Louisiana
  - AQX/CMX site, Troy, Michigan
  - AQX/CMX site, Garden City, New York
  - AQX/CMX Site, Winston-Salem, North Carolina
  - AQX/CMX site, Toledo, Ohio
  - AQX/CMX site, DeSoto, Texas
- Canada (17):
  - AQX/CMX site, Calgary, Alberta
  - AQX/CMX site, Kelowna, British Columbia
  - AQX/CMX Site, Vancouver, British Columbia
  - AQX/CMX site, Victoria, British Columbia
  - AQX/CMX site, Halifax, Nova Scotia
  - AQX/CMX site, Barrie, Ontario
  - AQX/CMX site, Brampton, Ontario
  - AQX/CMX site, Brantford, Ontario
  - AQX/CMX site, Burlington, Ontario
  - AQX/CMX site, Kingston, Ontario
  - AQX/CMX site, Kitchener, Ontario
  - AQX/CMX site, Oakville, Ontario
  - AQX/CMX site, Toronto, Ontario
  - Dr Lesley Carr, Toronto, Ontario
  - AQX/CMX site, Granby, Quebec
  - AQX/CMX site, Montreal, Quebec
  - AQX/CMX site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597
- See also: The Interstitial Cystitis Association (ICA) is the only nonprofit association dedicated solely to improving the quality of healthcare and lives of people living with interstitial cystitis (IC). — http://www.ichelp.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AQX-1125 | Placebo
Started | 37 | 32
Completed | 33 | 29
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AQX-1125 | Placebo | Total
Number analyzed (Participants) | 37 | 32 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 27 | 56
  >=65 years | 8 | 5 | 13
Sex/Gender, Customized [Number; unit: participants]
  Female | 37 | 32 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 32 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 31 | 30 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 20 | 44
  United States | 13 | 12 | 25
Weight [Mean (Standard Deviation); unit: kg] | 67.3 (12.40) | 76.5 (16.34) | 71.5 (14.98)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (4.71) | 29.1 (5.62) | 27.5 (5.31)
Duration of Diagnosis [Mean (Standard Deviation); unit: Months] | 63.5 (54.43) | 76.3 (57.28) | 69.4 (55.73)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Daily Bladder Pain Score (e-Diary)
Description: Change from baseline to week 6 in the average daily bladder pain score using a standardized 11-point numerical rating scale (NRS) recorded by e-diary. The 11-point NRS ranges from 0-10 with 0 indicating 'no pain' and 10 indicating 'worst pain'.
Time Frame: Baseline to Week 6
Population: The intent-to-treat analysis population (ITT) is the set of subjects who were randomized and received at least one dose of study medication.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 37 | 32
units on a scale
  Baseline | 6.4 (0.14) | 6.7 (0.18)
  Week 6: Change from Baseline | -2.4 (0.37) | -1.4 (0.32)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; A sample size of 28 subjects per group had 80% power to detect a 1.5-point difference in the change from baseline pain score between AQX-1125 and placebo assuming a between-subject SD of 2.0 and a 2-sided 5% significance level. Average daily pain scores were calculated using an average of up to the last 7 recordings within 9 days before each visit. Missing data, including premature discontinuation, was imputed using the LOCF approach for the primary efficacy end point of average daily pain score; Test type: Superiority or Other; p = 0.061, ANCOVA; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.1 to 0.0]

2. Secondary Outcome: Change From Baseline in the Maximum Daily Bladder Pain Score (e-Diary)
Description: Change from baseline to week 6 in the maximum daily bladder pain score using a standardized 11-point numerical rating scale (NRS) recorded by e-diary. The 11-point NRS ranges from 0-10 with 0 indicating 'no pain' and 10 indicating 'worst pain'.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 37 | 32
units on a scale
  Baseline | 7.6 (0.17) | 7.9 (0.19)
  Week 6: Change from Baseline | -2.6 (0.42) | -1.4 (0.35)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; E-diary maximum daily pain scores were calculated using an average of up to the last 7 recordings within 9 days before each visit. Missing data, including premature discontinuation, was imputed using the LOCF approach for the secondary efficacy variable of maximum daily pain score; Test type: Superiority or Other; p = 0.030, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.5 to -0.1]

3. Secondary Outcome: Change From Baseline in the Average Bladder Pain Score (Clinic)
Description: Change from baseline to week 6 in the average daily bladder pain score using a standardized 11-point numerical rating scale (NRS) recorded at study visit. The 11-point NRS ranges from 0-10 with 0 indicating 'no pain' and 10 indicating 'worst pain'.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 37 | 32
units on a scale
  Baseline | 6.7 (0.19) | 6.7 (0.20)
  Week 6: Change from Baseline | -2.6 (0.46) | -1.1 (0.40)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.008, ANCOVA; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.8 to -0.5]

4. Secondary Outcome: Change From Baseline in the Maximum Bladder Pain Score (Clinic)
Description: Change from baseline to week 6 in the maximum daily bladder pain score using a standardized 11-point numerical rating scale (NRS) recorded at study visits. The 11-point NRS ranges from 0-10 with 0 indicating 'no pain' and 10 indicating 'worst pain'.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 37 | 32
units on a scale
  Baseline | 8.1 (0.22) | 8.0 (0.23)
  Week 6: Change from Baseline | -2.8 (0.55) | -1.1 (0.50)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.028, ANCOVA; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.0 to -0.2]

5. Secondary Outcome: Bladder Pain/Interstitial Cystitis Symptom Score [BPIC-SS]
Description: Change in baseline to week 6 in the BPIC-SS participant reported questionnaire total score. The total BPIC-SS score ranges from 0-38, with a higher score indicative of worse symptoms. A score of 19 or more was considered to be discriminating between IC/BPS and overactive bladder at screening.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 37 | 32
units on a scale
  Baseline | 29.6 (0.59) | 31.6 (0.58)
  Week 6: Change from Baseline | -8.8 (1.37) | -4.0 (1.17)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.011, ANCOVA; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-9.5 to -1.3]

6. Secondary Outcome: O'Leary-Sant Interstitial Cystitis Symptom Index/Problem Index [ICSI/PI]
Description: Change from baseline to week 6 in the O'Leary Sant Symptom and Problem Index combined total scores. Both the ICSI and ICPI consist of 4 questions with responses for the ICSI rated on a scale of 0-5 (maximum score of 20, with a higher score indicating worse symptoms) and for the ICPI on a scale of 0-4 (maximum score of 16, with a higher score indicating worse symptoms). For the combined ICSI/PI the maximum score is 36, with a higher score indicating worse symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 37 | 32
units on a scale
  Baseline (ICSI/PI) | 27.3 (0.83) | 30.2 (0.78)
  Week 6: Change from Baseline (ICSI/PI) | -7.3 (1.25) | -3.0 (1.04)
  Baseline (ICSI) | 14.4 (0.48) | 16.1 (0.51)
  Week 6: Change from Baseline (ICSI) | -3.8 (0.62) | -1.4 (0.57)
  Baseline (ICPI) | 12.9 (0.39) | 14.1 (0.34)
  Week 6: Change from Baseline (ICPI) | -3.6 (0.69) | -1.6 (0.52)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.007, ANCOVA — ICSI/PI; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-8.8 to -1.4]
Statistical Analysis 2: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.005, ANCOVA — ICSI; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-4.6 to -0.9]
Statistical Analysis 3: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.014, ANCOVA — ICPI; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-4.5 to -0.5]

7. Secondary Outcome: Short Form 12 Version 2.0 Health Survey [SF-12v2] Questionnaire
Description: Change from baseline to week 6 in the SF-12v2 questionnaire. Two parameters, PCS (physical component summary) and MCS (mental component summary) were calculated. Both components scores range from 0 to 100 with higher scores indicating better Quality of Life.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 37 | 32
units on a scale
  Baseline (Mental Component) | 46.4 (1.34) | 41.3 (2.20)
  Week 6: Change from Baseline (Mental Component) | 0.5 (1.97) | 4.0 (1.67)
  Baseline (Physical Component) | 41.4 (1.42) | 36.1 (2.11)
  Week 6: Change from Baseline (Physical Component) | 3.8 (1.55) | 1.8 (1.22)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.592, ANCOVA — Mental Component; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-6.3 to 3.6]
Statistical Analysis 2: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.221, ANCOVA — Physical Component; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-1.6 to 6.7]

8. Secondary Outcome: Voiding Frequency as Recorded by Diary Over a 24 Hour Period
Description: For a 24-hour period (within 3 days of the subsequent visit), subjects recorded the frequency of each void prior to visit. The outcome measure was the change from baseline at week 6.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: number of voids
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 37 | 32
number of voids
  Baseline | 15.7 (1.21) | 16.8 (1.26)
  Week 6: Change from Baseline | -3.6 (1.05) | -0.8 (0.75)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Analyses of the secondary variable was based on observed data without imputation; Test type: Superiority or Other; p = 0.040, ANOVA; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-5.5 to -0.1]

9. Other Pre Specified Outcome: AQX-1125 Concentrations in Plasma and Urine (Trough Values)
Description: AQX-1125 Plasma and Urine Concentrations were measured at week 4 and week 6.
Time Frame: Week 4 and Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- AQX-1125: AQX-1125 Plasma and Urine Concentrations at Week 4 and 6
Arm/Group | AQX-1125
Number analyzed (Participants) | 37
ng/mL
  Plasma Week 4 | 252 (129)
  Plasma Week 6 | 225 (127)
  Urine Week 4 | 49,863 (40,630)
  Urine Week 6 | 33,396 (27,873)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing of informed consent until discharge from study at Week 10
Description: Adverse events were any unfavorable medical occurrence reported by the subject during the study. In addition, abnormal findings noted during the vital signs, ECG, physical or ophthalmology examinations deemed by the Investigator to be clinically significant were captured as adverse events.
Arm/Group | AQX-1125 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32
Other Adverse Events (participants affected / at risk) | 19/37 | 25/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AQX-1125 (N=37) | Placebo (N=32)
Abdominal discomfort or pain (upper/lower) (Gastrointestinal disorders) | 3 | 5
Diarrhea (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3
Edema (including peripheral) (General disorders) | 0 | 2
Sinusitis + vital sinusitis (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Increased blood pressure (Investigations) | 0 | 2
Headache (Nervous system disorders) | 0 | 2
Interstitial Cystitis (Renal and urinary disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1st publication to be a joint publication within 18 months of completion or termination of the trial at all sites. If not done the PI can publish separately, pending sponsor review 60 days prior to publication. PI agrees to remove sponsor confidential info. If sponsor identifies info it wishes to obtain IP protection for, PI agrees to remove sponsor identified info, or delay publication until the sponsor obtains IP protection and 120 calendar days from 1st submission for review to sponsor.